CLINICAL TRIAL: NCT00835432
Title: Prospective Clinical, Morphometric and Histological Study on Augmentation Using BoneCeramic as Bone Substitute in Combination With Either Cross-Linked or Non Cross-Linked Collagen Membrane in Dehiscent Type of Defects .
Brief Title: Morphometric, Clinical and Histological Study on One Stage Bone Augmentation Using BoneCeramic (BCP) and Collagen Membranes
Acronym: BCP+Collagen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Anton Friedmann, Department of Periodontology, Charité Center 3, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA/2/054
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Dehiscent Type of Alveolar Bone Defect; One Stage Bone Augmentation
Keywords: Lateral augmentation; GBR; BoneCeramic; collagen membrane; histomorphometry; morphometry; reentry; biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ossix — Test group
  Other Names: cross-linked collagen membrane barrier
Device: Biogide — controls
  Other Names: non cross-linked collagen membrane barrier

SUMMARY:
Prospective randomized assessment of alveolar ridge alterations after augmenting dehisced areas by applying principles of guided bone regeneration (GBR) subsequently to implant installation.

Ossix as cross-linked and BioGide as non cross-linked degradable collagen membranes, both used in combination with biphasic Calcium-Phosphate (BoneCeramic) as bone substitute. Clinical measurements and impressions from the sites of interest are to be taken at the stage of augmentation and 6 months after. At six months re-entry non-standardized biopsies from augmented sites will be taken to determine newly grown tissue in quality and quantity.

Due to different degradation characteristics of the two collagen membranes used as barrier, amount of newly formed mineralized tissue is suspected to vary in tests and controls, respectively.

ELIGIBILITY:
Inclusion Criteria:

* alveolar ridge deficiences after tooth loss

Exclusion Criteria:

* systemic disorders (diabetes mellitus, morbus crown, etc.)
* pregnancy or lactating period

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Alteration in width of alveolar bone at implant location after augmentation in mm | 6 months

SECONDARY OUTCOMES:
Histomorphometry in regard to areas occupied by bone to soft tissue to grafting material | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anton Friedmann, Dr., PhD, Principal Investigator — Department of Periodontology Charité Center3 CBF, Assmannshauser Str. 4-6, 14197 Berlin, Germany